CLINICAL TRIAL: NCT06389019
Title: Whole-slide Image and CT Radiomics Based Deep Learning System for Prognostication Prediction in Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Mingzhao Xiao (Other)
Responsible Party: Sponsor-Investigator, Mingzhao Xiao, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: BLCA_CMUFH; K2024-187-01 (Other: The First Affiliated Hospital of Chongqing Medical University)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
Keywords: deep learning; Radiomics; Histopathological tissue slides; Tomography
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BLCA: patients with bladder cancer who had surgery like radical cystectomy or transurethral resection of bladder tumour (TURBT).
  Interventions: Other: Deep learning system for prognostication prediction in bladder cancer

INTERVENTIONS:
Other: Deep learning system for prognostication prediction in bladder cancer — develop and validate a deep learning system for prognostication prediction in bladder cancer based on CT radiomics and whole slide images.

SUMMARY:
Bladder cancer (BLCA), with its diverse histopathological features and varying patient outcomes, poses significant challenges in diagnosis and prognosis. Postoperative survival stratification based on radiomics feature and whole slide image feature may be useful for treatment decisions to improve prognosis. In this research, we aim to develop a deep learning-based prognostic-stratification system for automatic prediction of overall and cancer-specific survival in patients with BLCA.

DETAILED DESCRIPTION:
Bladder cancer can be difficult to diagnose and predict outcomes for, as the disease can vary greatly between patients. This research aims to develop a new system that uses artificial intelligence to analyze patient information, including images from surgery and scans. This system could then automatically predict a patient's overall survival and how likely they are to survive specifically from bladder cancer. This information could be used by doctors to make better treatment decisions for each patient.

ELIGIBILITY:
Inclusion Criteria:

* patients with bladder cancer who had surgery like radical cystectomy or transurethral resection of bladder tumour (TURBT)
* contrast-CT scan less than two weeks before surgery
* complete CT image data and clinical data
* complete whole slide image data

Exclusion Criteria:

* patients with a postoperative diagnosis of non-urothelial carcinoma
* poor quality of CT images
* incomplete clinical and follow-up data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included patients who had surgery only or who had neoadjuvant chemotherapy before surgery. We excluded patients with a postoperative diagnosis of non-urothelial carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  the time from the date of surgery to death from any cause or the date of last contact (censored observation) at the date of data cut-off.

SECONDARY OUTCOMES:
Recurrence free survival | up to 10 years
  the time from the date of surgery to the date of first documented disease recurrence. Patients without recurrence at the time of analysis will be censored

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the current study are not publicly available due to the privacy of patients but are available from the corresponding author on reasonable request.